CLINICAL TRIAL: NCT04500106
Title: An Observational Study to Investigate the Feasibility and Patient/Caregiver/Investigator Satisfaction of Video-assisted Telenursing Use in Nurse Support Programs With LCIG
Brief Title: Study to Assess Participant/Caregiver/Investigator Satisfaction of Video-Assisted Telenursing in Adult Participants With Parkinson's Disease Treated With Levodopa-Carbidopa Intestinal Gel
Acronym: FACILITATECARE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-184
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Parkinson's Disease
Keywords: Levodopa-Carbidopa; LCIG; FACILITATE-CARE
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants With Nurse Support, Using Video Devices: Participants treated with Levodopa Carbidopa Intestinal Gel (LCIG) in accordance with approved label who are provided AbbVie Duodopa Specialist (ADS) nurse support, using video devices.
- Participants With Nurse Support, Not Using Video Devices: Participants treated with Levodopa Carbidopa Intestinal Gel (LCIG) in accordance with approved label who are provided AbbVie Duodopa Specialist (ADS) nurse support, not using video devices.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. The purpose of this study is to see how feasible and how satisfied participants/caregivers/investigators are with video-assisted telenursing use in nurse support programs with LCIG.

LCIG is an approved drug to treat PD. Approximately 50 adult participants with advanced PD will be enrolled in the study at approximately 10 sites across the world.

The study has 2 groups. In one group, around 25 participants will receive nurse support using video devices. In the second group, around 25 participants will receive nurse support without using video devices. All participants will attend a baseline visit and follow up visits at Week 4 and Week 12. The planned observation period will be 12 weeks.

Participants who are prescribed LCIG by their physicians will have three study related visits. Participants, caregivers, and investigators will be asked to complete questionnaires for the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Levodopa-Carbidopa Intestinal Gel (LCIG) therapy in accordance with the approved local LCIG label in the participating country
* Formerly LCIG-naive participants who have completed an in-hospital titration, have a Percutaneous Endoscopic transGastric Jejunostomy (PEG-J) placed and are discharged from hospital
* Decision to treat with LCIG made by the investigator prior to any decision to approach the participant to participate in this study
* Owns a telecommunication device equipped for videoconferencing (smart phone, tablet, laptop)
* Willing and able (based on investigator's judgment) to handle the video functionality of the device
* Caregiver willing to provide written informed consent

Exclusion Criteria:

* Any condition included in the contraindications section of the approved local LCIG label in the participating country
* Lack of caregiver support
* Participation in a concurrent interventional clinical trial
* Lack of motivation or insufficient language skills to complete the study questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with advanced Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Participant Acceptance of the AbbVie Duodopa Specialist (ADS) Nurse Support and Communication Access | At Week 12
  Participant acceptance is measured by the participant satisfaction with the AbbVie Duodopa Specialist (ADS) nurse support and communication access (Visual Analog Sore from 1 to 10).

SECONDARY OUTCOMES:
Participant Satisfaction With ADS Nurse Support and Communication Access | Through Week 12
  Participant Satisfaction is defined as participant satisfaction with the ADS nurse support and communication access at Week 4 (Visual Analog Scale [VAS] scoring from 1 to 10) and at Week 12 (VAS scoring from 8 to 10).
Participant Satisfaction with the ADS Nurse Support and Communication Access | At Week 12
  Participant satisfaction with the ADS nurse support and communication access is based on scoring 8 to 10 on a VAS (Binary: Yes/No).
Caregiver Satisfaction With ADS Nurse Support and Communication Access | Baseline (Week 0) to Week 12
  Caregiver satisfaction is measured as the satisfaction of caregiver with the ADS nurse support and communication access at weeks 4 and 12 (VAS from 1 to 10).
Caregiver Acceptance of ADS Nurse Support and Communication Access | Through Week 12
  Caregiver acceptance is measured as the acceptance of caregiver with the ADS nurse support and communication access at weeks 4 and 12 (VAS from 1 to 10).
Investigator Satisfaction With Nurse Support | At Week 12
  Investigator satisfaction is measured as the satisfaction of investigator with the nurse support (VAS from 1 to 10).
Participant Satisfaction With Video Functionality of the Device | Through Week 12
  Participant satisfaction is defined as the measure of satisfaction of participant with the video functionality of the device specifically at weeks 4 and 12 (VAS from 1 to 10).
Change of Caregiver Burden | Baseline (Week 0) to Week 12
  Change of caregiver burden will be measured by the Modified Caregiver Strain Index (MCSI). MCSI is a questionnaire comprising of 13 questions around major domains, to be filled by caregivers. The higher the score, the higher the level of caregiver strain. Scoring ranges from 0 to 26, with 0 indicating no strain and 26 indicating extreme strain.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Australia (3):
  - Royal Brisbane and Women's Hospital /ID# 223138, Herston, Queensland
  - Kingston Centre /ID# 222563, Cheltenham, Victoria
  - The Royal Melbourne Hospital /ID# 223005, Parkville, Victoria
- Israel (4):
  - Soroka University Medical Center /ID# 222754, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 222470, Ramat Gan, Tel Aviv
  - Kaplan Medical Center /ID# 222753, Rehovot
  - Tel Aviv Medical Center /ID# 222471, Tel Aviv
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego /ID# 222934, Wroclaw, Lower Silesian Voivodeship
  - Mazowiecki Szpital Brodnowski /ID# 222933, Warsaw, Masovian Voivodeship
  - COPERNICUS Podmiot Leczniczy Sp. z o.o. - Szpital sw. Wojciecha Adalberta /ID# 222932, Gdansk, Pomeranian Voivodeship
- Switzerland (3):
  - Luzerner Kantonsspital /ID# 223038, Lucerne, Canton of Lucerne
  - Kantonsspital St. Gallen /ID# 227012, Sankt Gallen, Canton of St. Gallen
  - Universitätsspital Zürich /ID# 223035, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gurevich T, Evans A, Hassin-Baer S, Kagi G, Koziorowski D, Roszmann A, Bergmann L, Parra Riaza JC, Sanchez-Solino O, Slawek J. Satisfaction with videoconferencing support for levodopa-carbidopa intestinal gel: An observational study. Digit Health. 2024 Aug 30;10:20552076241271847. doi: 10.1177/20552076241271847. eCollection 2024 Jan-Dec. PMID 39224799
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-184&Latitude=&Longitude=&LocationName=#additional-resources-section